CLINICAL TRIAL: NCT02208921
Title: An Observational, Cross Sectional Study to Assess the Prevalence of Chronic Kidney Disease in Type 2 Diabetes Patients in India
Brief Title: An Observational, Cross Sectional Study to Assess the Prevalence of Chronic Kidney Disease (CKD) in Type 2 Diabetes Patients
Acronym: START-INDIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00050; NIS-DIN-XXX-2014/1 (Other: AstraZeneca)
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- T2DM patients with Chronic Kidney Disease: T2DM patients with Chronic Kidney Disease

SUMMARY:
This non-interventional, multi-centric, cross-sectional study is aimed to determine the prevalence of Chronic Kidney Disease in Indian patients with Type 2 Diabetes (T2DM). 3000 patients will be enrolled from 30 investigative sites all over the country. Each investigative site will be expected to enrol 100 subjects. All the procedures will be completed in a single day.

DETAILED DESCRIPTION:
This is an observational, multicenter, cross-sectional study to be conducted at 30 sites in India. Endocrinologist/ Diabetologist from multiple private clinics will evaluate the Type 2 Diabetes patients. The study will be conducted over 9-10 months and will be started after obtaining written approval of Independent Ethics Committee (IEC) and written Informed consent of the patient. . Each investigative site will be expected to enrol 100 subjects. All the procedures will be completed in a single day.

ELIGIBILITY:
Inclusion Criteria:

1. Known cases of T2DM.
2. Male and female patients aged 18 years and above.
3. Must provide written Informed consent.

Exclusion Criteria:

1. Patients with known type-1 diabetes.
2. Patients with any form of acute kidney injury based on investigator's discretion.
3. Patients on maintenance dialysis or known renal transplant patients.
4. Patients who have participated in any interventional study within past 3 months prior to entry in this study.
5. Pregnant women.
6. Patients with symptomatic Urinary Tract Infection (UTI) or with history of hematuria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 3000 T2DM patients of either gender with age of 18 years and more will be enrolled in the study after the Informed Consent Process.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of T2DM patients with Chronic Kidney Disease (CKD) | 1 day
  The proportion of T2DM patients with CKD as per GFR (Glomerular Filtration Rate)criteria. GFR below 90 ml/min/1.73 m2 is defined as CKD. we will also classify CKD into various groups as per the KDIGO 2013.

SECONDARY OUTCOMES:
Frequency of T2DM patients in various stages of CKD | 1 day
  The proportion of T2DM patients with CKD as per GFR (Glomerular Filtration Rate)criteria. We will also classify CKD into various groups as per the KDIGO (KIDNEY DISEASE IMPROVING GLOBAL OUTCOMES) 2013.
Frequency of T2DM patients with CKD in patients with different duration of T2DM | 1 day
  The proportion of T2DM patients with CKD as per GFR (Glomerular Filtration Rate)criteria.we will also classify CKD into various groups as per the KDIGO 2013.
Frequency of patients with HbA1C less than 7% in T2DM patients with and without CKD | 1 day
  Frequency of patients with HbA1C (Glycated Haemoglobin) less than 7% in T2DM patients with and without CKD. we will correlate prevalence of CKD with HbA1C level.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prasanna Kumar K.M, DM, Study Chair — Endocrinology Center for Diabetes and Endocrine Care
Locations (18):
- India (18):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chandigarh
  - Research Site, Chennai
  - Research Site, Coimbatore
  - Research Site, Delhi
  - Research Site, Ghaziabad
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Karnāl
  - Research Site, Kolkata
  - Research Site, Ludhiana
  - Research Site, Mumbai
  - Research Site, Noida
  - Research Site, Pune
  - Research Site, Rohtak
  - Research Site, Trivandrum

REFERENCES:
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3100&filename=Synopsis.pdf